CLINICAL TRIAL: NCT05299866
Title: The Effect of Low-dose of S-ketamine Combined With Sufentanil for Postoperative Patient-controlled Intravenous Analgesia in Patients Following Cesarean Section
Brief Title: The Effect of S-ketamine Combined With Sufentanil for Postoperative Analgesia in Patients Following Cesarean Section
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ling Dong (Other)
Responsible Party: Sponsor-Investigator, Ling Dong, clinical professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YXLL-KY-2021(071)
Record Dates: First submitted 2022-02-26; First posted 2022-03-29 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: S-ketamine; Analgesia, Patient-Controlled; Cesarean Section
MeSH Terms: conditions — Agnosia | interventions — Esketamine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S-ketamine group (Experimental): The pump is established with S-ketamine 1mg/kg, sufentanil 2microgram/kg, andondansetron16mg, diluted with normal saline to 100 ml.
  Interventions: Drug: S-ketamine
- Control group (Placebo Comparator): The pump is established with sufentanil 2microgram/kg, andondansetron16mg, diluted with normal saline to 100 ml.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S-ketamine — After surgery, patient-controlled analgesia is provided. The pump is established with S-ketamine 1mg/kg, sufentanil 2microgram/kg, andondansetron16mg, diluted with normal saline to 100 ml. The pump is programmed to deliver 2 ml boluses with a background infusion rate at 2 ml /h and a 30 min lockout interval.
  Arms: S-ketamine group
Drug: Placebo — After surgery, patient-controlled analgesia is provided. The pump is established with sufentanil 2microgram/kg, andondansetron16mg, diluted with normal saline to 100 ml. The pump is programmed to deliver 2 ml boluses with a background infusion rate at 2 ml /h and a 30 min lockout interval.
  Arms: Control group

SUMMARY:
This randomized controlled trial is designed to investigate the effect of low-dose of S-ketamine combined with sufentanil for postoperative patient-controlled intravenous analgesia in patients following cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status II
* Patients aged between 20 and 40 years
* 18 kg/m² ≤BMI≤30 kg/m²
* singleton term pregnancy
* scheduled for elective cesarean section

Exclusion Criteria:

* Refused to participant in this trial
* Severe heart dysfunction or pulmonary insufficiency
* Poor blood pressure control in those with hypertension (BP >160/100 mmHg in the ward)
* Previous history of Intracranial hypertension or hyperthyroidism
* Previous history of schizophrenia, epilepsy, myasthenia gravis or delirium
* Allergy to drugs used in the study

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Estimated)
Dates: Start 2022-04-12 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with moderate-to-severe pain | Up to 48 hours after surgery
  Moderate-to-severe pain is defined as a numeric rating scale (NRS; an 11-point scale where 0=no pain and 10=the worst pain) pain score ≥4.

SECONDARY OUTCOMES:
NRS pain score at rest and with movement | Hour 12 & Hour 24 & Hour 48 after surgery
  Pain is assessed with a numeric rating scale (NRS; an 11-point scale where 0=no pain and 10=the worst pain)

OTHER OUTCOMES:
The total number of presses of Patient-controlled Analgesia (PCA) | Up to 48 hours after surgery
  The total number of presses of PCA
The percentage of using rescue analgesics | Up to 48 hours after surgery
  The percentage of using rescue analgesics
The Richmond Agitation-Sedation Scale(RASS) | Hour 12 & Hour 24 & Hour 48 after surgery
  Sedation is assessed with a numeric rating scale(RASS;an 10-point scale with -5 to +4)
The incidence of postoperative adverse event | Up to 48 hours after surgery
  postoperative adverse event with nausea,vomiting,dizziness,nightmares, hallucination and etc

CONTACTS AND LOCATIONS:
Locations (1):
- Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brinck EC, Tiippana E, Heesen M, Bell RF, Straube S, Moore RA, Kontinen V. Perioperative intravenous ketamine for acute postoperative pain in adults. Cochrane Database Syst Rev. 2018 Dec 20;12(12):CD012033. doi: 10.1002/14651858.CD012033.pub4. PMID 30570761
- [Background] Schwenk ES, Viscusi ER, Buvanendran A, Hurley RW, Wasan AD, Narouze S, Bhatia A, Davis FN, Hooten WM, Cohen SP. Consensus Guidelines on the Use of Intravenous Ketamine Infusions for Acute Pain Management From the American Society of Regional Anesthesia and Pain Medicine, the American Academy of Pain Medicine, and the American Society of Anesthesiologists. Reg Anesth Pain Med. 2018 Jul;43(5):456-466. doi: 10.1097/AAP.0000000000000806. PMID 29870457
- [Background] Isik Y, Dag ZO, Tulmac OB, Pek E. Early postpartum lactation effects of cesarean and vaginal birth. Ginekol Pol. 2016;87(6):426-30. doi: 10.5603/GP.2016.0020. PMID 27418219
- [Background] Hobbs AJ, Mannion CA, McDonald SW, Brockway M, Tough SC. The impact of caesarean section on breastfeeding initiation, duration and difficulties in the first four months postpartum. BMC Pregnancy Childbirth. 2016 Apr 26;16:90. doi: 10.1186/s12884-016-0876-1. PMID 27118118